CLINICAL TRIAL: NCT01491542
Title: A Pilot Prospective Randomized Clinical Investigation of INFUSE® Bone Graft and MASTERGRAFT® Granules With the CD HORIZON® Spinal System for Posterolateral Lumbar Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: INFUSE® Bone Graft and MASTERGRAFT® Granules With CD HORIZON® for Posterolateral Lumbar Fusion in Patients With Degenerative Disc Disease - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-11
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: Symptomatic Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBMP-2 / ACS (Experimental)
  Interventions: Device: INFUSE® Bone Graft/MASTERGRAFT® Granules/CD HORIZON®
- Autogenous bone (Active Comparator)
  Interventions: Device: Autogenous Bone / CD HORIZON® Spinal System

INTERVENTIONS:
Device: INFUSE® Bone Graft/MASTERGRAFT® Granules/CD HORIZON® — The INFUSE® Bone Graft component of the investigational device consists of recombinant human Bone Morphogenetic Protein-2(rhBMP-2) and an absorbable collagen sponge (ACS)carrier. The MASTERGRAFT® Granules will be used as a type of bulking agent to provide compression resistance.
  Other Names: Infused Bone Graft; MasterGraft
  Arms: rhBMP-2 / ACS
Device: Autogenous Bone / CD HORIZON® Spinal System — The control will be autogenous bone taken from the iliac crest of the patient and placed bilaterally across two adjacent transverse processes and used in conjunction with the CD HORIZON® Spinal System.
  Other Names: Autograft
  Arms: Autogenous bone

SUMMARY:
The purpose of this pilot clinical trial is to evaluate the feasibility of using the investigational implant (INFUSE® Bone Graft and MASTERGRAFT® Granules with the CD HORIZON® Spinal System) as a method of facilitating spinal fusion in patients with symptomatic degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history (e.g., pain [leg, back, or symptoms in the sciatic nerve distribution], functional deficit and/or neurological deficit) and radiographic studies (e.g.,C T, MRl, X-Ray,etc.) to include one or more of the following:

   * instability (defined as angulation ≥ 5° and/or translation ≥ 4mm,based on flexion/extension radiographs);
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score ≥ 30.
3. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding HW,1932).
4. Requires fusion of a single level disc space from L1 to S1.
5. Is at least 18 years of age, inclusive, at the time of surgery.
6. Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of 6 months.
7. If of child-bearing potential, patient is non-pregnant,non-nursing,and agrees to use adequate contraception for 1 year following surgery.
8. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Has primary diagnosis of a spinal disorder other than degenerative disc disease with Grade 1 or less spondylolisthesis at the involved level.
2. Had previous spinal fusion surgical procedure at the involved level or an adjacent level.
3. Requires spinal fusion at more than one lumbar level.
4. Has a condition which requires postoperative medications that interfere with fusion, such as steroids or prolonged use of nonsteroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
5. Has a documented history of osteopenia or osteomalacia.
6. Has any of the following that may be associated with diagnosis of osteoporosis (if "Yes" to any of the below risk factors,a dual x-ray absorptiometry (DEXA) scan will be required to determine eligibility.)

   * Postmenopausal non-black female over 60 years of age and weighs less than 140 pounds.
   * Postmenopausal female that has sustained a non-traumatic hip, spine, or wrist fracture.
   * Male over the age of 70.
   * Male over the age of 60 that has sustained a non-traumatic hip or spine fracture. If the level of BMD is a T score of -3.5 or a T score of -2.5 with vertebral crush fracture,then the patient is excluded from the study.
7. Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
8. Has overt or active bacterial infection, either local or systemic.
9. Has a documented titanium alloy allergy or intolerance.
10. Is mentally incompetent. If questionable, obtain psychiatric consult.
11. Has a 'Waddell Signs of Inorganic Behavior'score of 3 or greater.
12. Is a prisoner.
13. Is an alcohol and/or drug abuser as defined by currently undergoing treatment or alcohol and/or drug abuse.
14. ls a tobacco user at the time of surgery.
15. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate).
16. Has a documented history of autoimmune disease ( e.g. Systemic Lupus Erythematosus or dermatomyositis).
17. Has a history of exposure to implanted collagen or silicone implants.
18. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
19. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS/MASTERGRAFT® Granules implantation.
20. Has received any previous exposure to any/all BMP's of either human or animal extraction.
21. Has a history of allergy to bovine products or a history of anaphylaxis.
22. Has a history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease,renal osteodystrophy, Ehlers- Danlos syndrome,or osteogenesis imperfecta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-04; Primary Completion 2006-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Overall Success | 24 months
  A patient will be considered an overall success if all of the following conditions are met:
  1. Fusion;
  2. Postoperative Oswestry score improvement of at least 15% from preoperative;
  3. Maintenance or improvement in neurological status;
  4. No serious adverse event classified as implant associated or implant surgical procedure associated;
  5. No additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
General Health Status (SF-36) | 24 months
Pain Status (back pain, leg pain) | 24 months
Patient Satisfaction | 24 months
Patient Global Perceived Effect | 24 months